CLINICAL TRIAL: NCT05538949
Title: A Phase I Clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetics of EB-203 Eye Drops in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of EB-203 Eye Drops in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EyebioKorea, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB-203-101
Record Dates: First submitted 2022-08-29; First posted 2022-09-14 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Participants received 1%, 2%, 4%, 8% of EB-203 eye drops. Group A : EB-203 1% eye drops, Group B : EB-203 2% eye drops, Group C : EB-203 4% eye drops, Group D : EB-203 8% eye drops
  Interventions: Drug: EB-203
- Placebo group (Placebo Comparator): Participants received Placebo eye drops. Group A : Placebo eye drops, Group B : Placebo eye drops, Group C : Placebo eye drops, Group D : Placebo eye drops
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EB-203 — * Single dose : EB-203 1%, 2%, 4%, 8% 1Drop, QD / Day1.
  * Multiple dose : EB-203 1%, 2%, 4%, 8% 1Drop, BID / Day5~Day8.
  Arms: Test group
Drug: Placebo — Placebo 1Drop, QD / Day1, BID / Day5~Day8.
  Arms: Placebo group

SUMMARY:
The purpose of study is to evaluate safety, tolerability and pharmacokinetics of EB-203 Drops in adult healthy volunteers.

condition/disease : AMD(Age-related Macular Degeneration) Intervention/treatment : EB-203 or Placebo Phase : Phase I

DETAILED DESCRIPTION:
Study Title : A Phase I clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetics of EB-203 Eye Drops in Healthy Volunteers

Purpose : The purpose of study is to evaluate safety, tolerability and pharmacokinetics of EB-203 Drops in adult healthy volunteers

Number of Site : One site (INJE UNIVERSITY BUSAN PAIK HOSPITAL)

A total of 8 subjects will be dosed in each group(Group B, C, D) with subjects randomized 3:1 to EB-203 or placebo.(A total of 4 subjucts will be dosed in Group A) Up to 28 subjects will be enrolled in four consecutive cohorts. A safety data review as masking will be performed for 4days prior repeated treatment. Treatment of high dose will proceed following a review of safety data from low dose.

Safety and tolerability assessments and drug plasma concentrations will be evaluated throughout the study in all cohorts.

Outcome Measures :

1. Primary Outcome Measures

   : Frequency of AEs (Adverse Events) and ADR (Adverse Drug Reaction)
2. Secondary Outcome Measures : Pharmacokinetic variables evaluation for single and repeated dose administration.

Safety Assessment :

* V/S, Physical Exam, Laboratory Exam, ECG
* Ophthalmic Exam

Investigational product(IP) :

* Active Comparator : 1 %, 2 %, 4 %, 8% of EB-203
* Placebo Comparator : Placebo

Intervention&Number of Subject : Total 28 subjects (A Group 4, B~D Group 8)

Inclusion Criteria :

1. Healthy adult males between the ages of 20 and 55 years
2. Body Weight > 55 kg and BMI 18 ~ 27 kg/m2
3. Patients signed informed consent willing and able to sign informed consent form and comply with visit and study procedures per protocol

Exclusion Criteria :

1. A person who has a history or presence of clinical significant Cardiovascular, Respiratory, Hepatobiliary, Renal/Urinary, Hematological, Gastrointestinal, Endocrine, Neurological, Psychiatric disease
2. A person who has the following diseases from medical and ophthalmic examination

   * Suspected symptoms or signs of visual organ disease including corneitis, uveitis, retinitis, dry eyes, and strabismus
   * Corrected visual acuity < 20/25 or Intraocular Pressure > 21 mmHg
   * Patients who have received any eye surgery
   * Other abnormal findings in ophthalmic examinations
3. Other patients considered by investigators to be inappropriate as subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males between the ages of 20 and 55 years
* Body Weight > 55 kg and BMI 18 ~ 27 kg/m2
* Patients signed informed consent willing and able to sign informed consent form and comply with visit and study procedures per protocol

Exclusion Criteria:

* A person who has a history or presence of clinical significant Cardiovascular, Respiratory, Hepatobiliary, Renal/Urinary, Hematological, Gastrointestinal, Endocrine, Neurological, Psychiatric disease
* A person who has the following diseases from medical and ophthalmic examination

  * Suspected symptoms or signs of visual organ disease including corneitis, uveitis, retinitis, dry eyes, and strabismus
  * Corrected visual acuity < 20/25 or Intraocular Pressure > 21 mmHg
  * Patients who have received any eye surgery
  * Other abnormal findings in ophthalmic examinations
* Other patients considered by investigators to be inappropriate as subjects.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Frequency of AEs (Adverse Events) and ADR (Adverse Drug Reaction) | Single dose : up to 4 Days, Multiple dose : up to Day10, PSV
  V/S, Physical Exam, ECG, Laboratory Exam, Ophthalmic Exam

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Day1, Day2, Day8, Day9, Day10
  Cmax of EB-203 was derived across all post-dose PK collections and expressed in μg/mL.
Area under the plasma concentration versus time curve (AUC) | Day1, Day2, Day8, Day9, Day10
  AUC of EB-203 in serum over the time interval from 0 extrapolated to infinity. Values for AUC of EB-203 were expressed in days by micrograms per milliliter (days•μg/mL).
Time to Maximum Serum Concentration (Tmax) | Day1, Day2, Day8, Day9, Day10
  Tmax of EB-203 was based on the Cmax derived across all post-dose PK collections and expressed in hours.
Terminal Elimination Half-Life (T1/2) | Day8.
  T1/2 of EB-2-3 was derived across all PK collections and expressed in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Lyul Ghim, Principal Investigator — Busan Paik Hospital, Inje University
Locations (1):
- Busan Paik Hospital, Inje University, Busan, South Korea